CLINICAL TRIAL: NCT03569254
Title: Effectiveness, Safety and Perceptions With the Use of One LED Blanket Device in the Ambulatory Treatment of Neonatal Jaundice
Brief Title: Effectiveness, Safety and Perceptions With the Use of One LED Blanket Device in the Ambulatory Treatment of Jaundice
Acronym: LEDlightT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathalie Charpak (Other)
Collaborators: Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor-Investigator, Nathalie Charpak, Director, Kangaroo Foundation
Organization: Kangaroo Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/187
Record Dates: First submitted 2018-06-04; First posted 2018-06-26 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Jaundice, Neonatal; Phototherapy
Keywords: infant, newborn; devices; treatment; hyperbilirubinemia
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Intervention Model Description: Parallel assignment randomized controlled clinical trial with preterm or low birth weight infants who have low risk hyperbilirubinemia requiring phototherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neomedlight Phototherapy Blanket (Experimental): Phototherapy with a fiber-optic device based on LED light administered intermittently for a total of 6 hours with periods of 2 hours in kangaroo position and pauses of 1 hour at the end of each period.
  Interventions: Device: Neomedlight Phototherapy Blanket
- Ohmeda-Fiber Optic Phototherapy Blanket (Active Comparator): Phototherapy with a fiber-optic device: the Ohmeda fiber optic Phototherapy blanket
  Interventions: Device: Ohmeda-Fiber Optic Phototherapy Blanket

INTERVENTIONS:
Device: Neomedlight Phototherapy Blanket — The NeoMedLight® phototherapy blanket is an innovative new fiber-optic device based on LED light. Its light emitting surface area is 40.5x30 cm or 1200 cm2. The device size is 40.5 x30 cm. It incorporates fiber optic mesh and is protected by a vinyl cover and a disposable liner for patient comfort and hygiene. This device provides therapeutic light (404-515nm) to a wide extension of the body surface area. Its average irradiation footprint is 35uW / cm2 / nm ± 15%. The phototherapy was done intermittently in periods of 2 hours with 1 hour of rest for a total time of 6 hours in kangaroo position.
  Arms: Neomedlight Phototherapy Blanket
Device: Ohmeda-Fiber Optic Phototherapy Blanket — This device is a high performance version of Ohmeda Medical's Biliblanket that uses a fiber optic cable to deliver light from a high-intensity lamp to a device composed of a fiber optic fabric. The device has a disposable liner and is left in direct contact with the patient. The patient is exposed to a light with a wavelength between 400 and 550 nanometers. The phototherapy system consists of a light emitting unit, a fiber optic cable four feet long (121.9 cm) and a lightweight mattress. It has two available sizes: 4.38 x 9.38 inches (11.12 x 23.83 cm) and 4.00 x 6.00 inches (10.16 x 15.2 cm).
  Arms: Ohmeda-Fiber Optic Phototherapy Blanket

SUMMARY:
Objective: to evaluate the effectiveness, safety and level of satisfaction of parents and healthcare team with one innovative device for phototherapy to which a LED light mesh has been incorporated(a blanket), comparing it with the Ohmeda BiliBlanket Plus®. Methods: randomized controlled clinical trial with preterm or low birth weight infants requiring phototherapy. The study protocol was evaluated and accepted by the San Ignacio Hospital and "Pontificia Universidad Javeriana" research committee. Informed consent was requested from parents and the authors declared no conflict of interest. Sample size and allocation: using the STATA 12 program, a sample size of 64 patients was calculated(5% losses), 32 for each group, with significance level of 0.05, power of 80% and difference in bilirubin decreasing of at least 0,1 mg/dl/h with standard deviation of 0.14 mg/dl/h. A computer program randomized the allocation to the intervention and the concealment of the assignment was through sealed opaque envelopes. Seric bilirubin levels were taken at the start and at the end of phototherapy. Controls were done every 2 hours with the Bilicheck spectrophotometer device. Axillary temperature was measured at the beginning of phototherapy, at 30 min, 60 min, and every 2 hours during intervention. Physical examination and recording of side effects related were performed. Parents and health personnel answered a survey on comfort and perceptions with the use of the devices at the end of phototherapy. Analysis: Comparison of means was made for the decrease of bilirubin levels and body temperatures and chi-square for incidence of side effects and results of the survey.

DETAILED DESCRIPTION:
Background: Jaundice due to hyperbilirubinemia is the most common entity that requires medical management in neonates. About 50% of full-term newborns and 80% of premature infants develop jaundice. The effectiveness of phototherapy for neonatal jaundice depends on two factors: the spectrum of light emitted and the spectral irradiation of light. An ideal phototherapy device should have a broad light emission surface, in order to cover the maximum of the body surface in the horizontal plane, it should be durable, generate relatively little heat and provide a wavelength and light intensity (radiation) optimal (460-490nm and ≥ 30uw / cm2 / nm). The conventional phototherapy devices use fluorescent lamps that emit heat and require eye protectors, in addition to increasing water losses, which requires a permanent monitoring of vital functions and temperature. Its use imposes hospitalization and consequently mother-child separation, always traumatic. The most recent devices use light emitting diodes (LED light) as the light source. Objective: to evaluate the effectiveness, safety and level of satisfaction of parents and healthcare team with one innovative device for phototherapy to which a LED light mesh has been incorporated (one blanket), comparing it with the Ohmeda BiliBlanket Plus®, used at the Kangaroo Mother Care Program for intermittent ambulatory phototherapy. Methods: randomized controlled clinical trial with preterm or low birth weight infants that required phototherapy according to the guidelines of the American Academy of Pediatrics. The Protocol was evaluated and accepted by the "Hospital Universitario San Ignacio and Pontificia Universidad Javeriana research committee". Informed consent was requested from parents and the authors declared no conflict of interest. Sample size and allocation: using the STATA 12 program, a sample size of 64 patients was calculated, 32 for each group, with significance level of 0.05, power of 80% and difference in bilirubin decreasing of at least 0,1 mg/dl/h with standard deviation of 0.14 mg/dl/h and 5% of losses. A computer program randomized the allocation to the intervention and the concealment of the assignment was through sealed opaque envelopes. Seric bilirubin levels were taken at the start and at the end of phototherapy. Controls were done every 2 hours with bilicheck spectrophotometer device. Axillary temperature was measured at the beginning of phototherapy, at 30 min, 60 min, and every 2 hours during intervention. Physical examination, recording of side effects related, mortality and requirement of hospital treatment were performed. Parents and health personnel answered a survey on comfort and perceptions with the use of the devices at the end of phototherapy. Analysis: Comparison of means was made for the decrease of bilirubin levels and body temperatures and chi-square for incidence of side effects, hospitalization, mortality and results of the survey.

ELIGIBILITY:
Inclusion Criteria:

* Low Risk Hyperbilirubinemia requiring phototherapy according to the guidelines of the American Academy of Pediatrics and recommendations for management of premature infants under 35 weeks, adopted by the Kangaroo Mother Care Ambulatory Program.
* Start of jaundice at a chronological age greater than 48 hours.
* Bilirubin level ≤18 mg / dL
* Knowledge of blood groups of mother and child.
* Parents are required to sign informed consent where they agree to participate in the study.

Exclusion Criteria:

* Parents without availability to stay in the Kangaroo Mother Care Program for at least 6 hours.
* Extensive skin lesions due to burns or sloughing at the physical examination prior to entering the study.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Bilirubin change rate in mg/dl/h | through study completion, an average of 6 hours
  Bilirubin lowering rate (initial seric bilirubin- final seric bilirubin/time of phototherapy).

SECONDARY OUTCOMES:
Patient temperature during phototherapy | through study completion, an average of 6 hours
  Axillary temperatures at 30 min, 60 min, 1 hour, 2 hours, 4 hours and 6 hours of phototherapy.
Incidence of skin lesions related to phototherapy | through study completion, an average of 6 hours
  rash, burns, etc... related to phototherapy
Incidence of dehydration related to phototherapy | through study completion, an average of 6 hours
  Dehydration documented with physical examination and weight
Incidence of diarrhea related to phototherapy | through study completion, an average of 6 hours
  Documented diarrhea
Incidence of other side effects related to phototherapy | through study completion, an average of 6 hours
  Other effects recorded in clinic history related to phototherapy
Perceptions of parents with the use of devices | At study completion, an average of 6 hours.
  Comfort with heat, humidity, breastfeeding, proximity and possibility of contact with the baby. The investigators did a validated survey at the end of treatment using a Likert scale(1-7): 1=uncomfortable. 7=comfortable. 4=indifferent
Perceptions of the health team with the use of the devices | At study completion, an average of 6 hours.
  Comfort cleaning and using the device and comfort with light, heat, humidity, and feeding and taking care of the baby. The investigators did a validated survey at the end of treatment using a Likert scale(1-7): 1=uncomfortable. 7=comfortable, 4=indifferent
Hospitalization for hyperbilirubinemia | Between beginning of treatment and 72 hours after
  Rate of hospitalization for hyperbilirubinemia
Mortality | Between beginning of treatment and 72 hours after
  Rate of mortality related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Charpak, Dr., Study Director — Kangaroo Foundation Director
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No